CLINICAL TRIAL: NCT04301427
Title: Smallest Significant Value in Osteodensitomery in an Obese Population
Acronym: PPVS-ob
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO20019
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: Bone density; Osteoporosis; Osteopenia; Obesity; OSteodensitometry
MeSH Terms: conditions — Obesity; Osteoporosis; Bone Diseases, Metabolic | interventions — Bone Density

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese patient (Other)
  Interventions: Other: Bone mineral density

INTERVENTIONS:
Other: Bone mineral density — Bone mineral density will be measured twice in all included patients.

SUMMARY:
The aim of this study is to determined the smallest significant value in osteodensitometry in obese population. The study population will be divided in 3 groups according to their BMI.

Bone mineral density will be measured twice in osteodensitometry, then the smallest significant value will be determined.

Our hypothesis is that the smallest significant value that we use in an non-obese population can be different in an obese population.

DETAILED DESCRIPTION:
The aim of this study is to determined the smallest significant value in osteodensitometry in obese population.

There will be at least 120 patient included. The study population will be divided in 3 groups according to their BMI : the first group has a BMI between 30 and 35 kg/cm² ; the second group has a BMI between 35 et 40 kg/cm² ; and the third group has a BMI over 40 kg/cm².

Patients will be referred by their doctors (rheumatologist and others) to evaluate their bone mineral density in osteodensitometry at CHU of Reims. Patients will be informed of the aim of the study by the prescriptor of the osteodensitometry.

The osteodensitometry will be executed by a nurse. Patients will have to complete a questionnaire about their medical history and their medications.

Bone mineral density will be measured twice in osteodensitometry, at the lumbar spine, the hip and the femur. This exam lasts approximately 40 minutes.

Then the smallest significant value will be determined by comparing each measure for every patients.

ELIGIBILITY:
Inclusion criteria :

* Major patients
* Patients referred to the CHU of Reims to make an osteodensitometric evaluation of their bone mineral density
* BMI > 30 kg/cm²
* Patient affiliated to a health insurance plan
* Patients who have signed informed consent

Exclusion criteria :

* Minor patients
* Pregnant women
* Patients protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
osteodensitometry in obese population | Day 1
  smallest significant value in osteodensitometry in obese population

SECONDARY OUTCOMES:
osteodensitometry in obese population with BMI between 30 and 35 kg/cm² | Day 1
  smallest significant value in osteodensitometry in obese population with BMI between 30 et 35 kg/cm²
osteodensitometry in obese population with BMI between 35 and 40 kg/cm² | Day 1
  smallest significant value in osteodensitometry in obese population with BMI between 35 et 40 kg/cm²
osteodensitometry in obese population with BMI over 40 kg/cm² | Day 1
  Smallest significant value in osteodensitometry in obese population with BMI over 40 kg/cm²

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Dorilleau C, Kanagaratnam L, Charlot I, Hittinger A, Bertin E, Salmon JH, Geoffroy M. "The least significant change on bone mineral density scan increased in patients with higher degrees of obesity". Aging Clin Exp Res. 2024 Apr 23;36(1):98. doi: 10.1007/s40520-024-02736-4. PMID 38652346